CLINICAL TRIAL: NCT04530149
Title: Vital Capacity in Ultrasound Guided Serratus Plane Block in Emergency Department Patients With Multiple Rib Fractures: A Randomized Controlled Trial
Brief Title: Vital Capacity in Ultrasound Guided Serratus Plane Block in ED Patients With Multiple Rib Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The original PI left the institution; COVID interrupted the study; difficult enrolling patients.
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-03-17
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: Pain; Pain management; Rib
MeSH Terms: conditions — Pain; Agnosia | interventions — Acetaminophen; Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- serratus anterior plane block group (Active Comparator): The injection of bupivicaine into the chest muscle is performed with an ultrasound machine which can see the needle as it enters the muscle. The skin is cleaned with a sterile solution and the needle is guided right next to the chest muscle where either the bupivicaine injected. After the injection, the needle is taken out.
  Interventions: Drug: Acetaminophen; Drug: Bupivacain
- Placebo injection group (Placebo Comparator): The injection of normal saline into the chest muscle is performed with an ultrasound machine which can see the needle as it enters the muscle. The skin is cleaned with a sterile solution and the needle is guided right next to the chest muscle where saline is injected. After the injection, the needle is taken out.
  Interventions: Drug: Acetaminophen; Drug: Saline

INTERVENTIONS:
Drug: Acetaminophen — receive ketamine 0.15 mg/kg IV in 100 mL normal saline over 30 minutes for pain
Drug: Bupivacain — The injection of bupivicaine into the chest muscle is performed with an ultrasound machine which can see the needle as it enters the muscle.
  Arms: serratus anterior plane block group
Drug: Saline — The injection of saline into the chest muscle is performed with an ultrasound machine which can see the needle as it enters the muscle.
  Arms: Placebo injection group

SUMMARY:
I. Background:

Patients with multiple rib fractures are challenging from both pulmonary and analgesia perspectives. Adequate pain management is essential in prevention of complications secondary to decreased inspiratory volume. Significant morbidity and mortality of rib fractures is secondary to severe pain that limits ribcage movement, decreases inspiratory volumes and causes inadequate cough. Decreased vital capacity predisposes patients to atelectasis, abnormal mucous clearance and pneumonia. The objective of this study is to assess the efficacy of the serratus anterior plane block (SAPB) in improvement of vital capacity in patients with multiple unilateral rib fractures when compared to conventional management with medications. Currently, evidence of efficacy of SAPB in managing pain secondary to multiple rib fractures is limited to case reports and series, none of which evaluate vital capacity.

II. Significance:

The findings of this study may indicate that SAPB is superior to pharmacological management in increasing vital capacity in patients with multiple unilateral rib fractures and suggest SAPB for first line therapy in patients with rib fractures. The findings may decrease the risk of pulmonary complications as well as the use of opiates in management of multiple rib fractures in the Emergency Department especially in patients with numerous comorbidities and contraindications to conventional treatment modalities. This study may support the need for training emergency medicine physicians in bedside SAPB in order to provide the optimal therapy for patient with multiple unilateral rib fractures.

III. Study Objectives:

The primary objectives are to evaluate whether ultrasound guided SAPB results in a greater improvement in percent predicted vital capacity compared to standard therapy with a sham injection. The investigators will also evaluate pain scores and the safety profile of the SAPB procedure compared to those receiving standard analgesia.

IV. Hypothesis:

The primary hypothesis is that SAPB is superior to sham injection in improving the percent of predicted vital capacity. The secondary hypothesis is that SAPB will have greater improvement in pain scores and have a superior safety profile compared to placebo injection.

DETAILED DESCRIPTION:
STUDY DESIGN

This is a single center prospective, randomized, blinded clinical trial with a convenience sample that will be conducted in the Emergency Department of an urban level I trauma center.

A. Identify and enroll all patients coming in to the ED patient with presumed or clinically apparent 2 or more unilateral rib fractures between T3 to T9, with a resting pain score of ≥5. All patients meeting exclusion criteria will be excluded.

B. Randomization procedure:

1. Pharmacy will dispense 30mL of injectate which will be randomized in block of 10 to either the SAPB group (30mL of 0.25% bupivacaine with epinephrine) or sham group (30mL of normal saline).

C. Injection

1. Patient consent will be obtained and time out will be performed on all patients.
2. Patients will be placed on cardiac monitor and placed in lateral decubitus or if unable to turn, they will be supine.
3. Under the usual sterile technique, the serratus anterior muscle overlying the 5th rib at the mid-axillary line will be identified with ultrasound.
4. A spinal needle will be introduced in-plane under ultrasound guidance and advanced until the needle tip is located in the fascial plane just above the serratus anterior muscle. The needle tip will not be advanced unless completely visualized under ultrasound.
5. Normal saline will be injected first to determine correct location of the needle tip. Spreading of fluid along the fascial plane will confirm the correct location of the needle tip.
6. The normal saline will then be switched to the study drug of which 30mL of either normal saline or 0.25% bupivacaine with epinephrine which will then be injected into the fascial plane as described in Blanco et al, and Hetta et al.
7. The study drug will be injected 5mL at a time and the patient will be asked if any symptoms of Local Anesthetic Systemic Toxicity (LAST toxicity) are present (perioral numbness, tinnitus, dizziness).
8. After injection is completed the needle will be withdrawn and patient will remain on the cardiac monitor for another 30 minutes to monitor for symptoms of LAST toxicity (Di Gregorio).
9. This procedure was based on the serratus anterior plane block protocol from Khalil et al.

D. Slow Vital Capacity (SVC) Measurement

1. SVC will be performed using spirometer that has been internally validated
2. SVC will be performed by physicians trained by the respiratory therapy department and who have demonstrated validation compared to respiratory therapist obtained SVC values
3. The patient will be sitting up when performing SVC and a script will be followed as to how to educate and coach the patient on performing appropriate incentive spirometry technique.
4. At least 3 SVC measurements within 150mL of each other are required to qualify for an accurate measurement.
5. The maximum of these 3 SVC values and a corresponding % predicted SVC will be obtained and considered the maximum % predicted SVC.
6. % Predicted SVC will be obtained based on the National Health and Nutrition Examination Survey (NHANES III) calculator through the CDC.

E. Pain scores

1. Subjects will be asked to rate their maximum pain score from 0-10 with resting breathing and with deep breaths.

Design:

A. Potential study patients will be identified through review of the emergency department (ED) electronic board, and ED physicians will also screen for potential study patients. Pain scores are assessed in triage as is standard in the ED.

B. If the patient has pain from presumed or clinically apparent 2 or more unilateral rib fractures between T3 to T9, and he/she has a resting pain score of ≥5 on the Numeric Pain Rating Scale, where 0 is no pain, 5 is moderate pain, and 10 is the worst possible pain upon initial assessment, then he/she will be eligible to participate in the study.

The patient will then be asked to participate if he/she does not have any exclusion criteria.

C. At time of enrollment, the patient will have recorded pain scores, vital signs, and slow vital capacity measured.

D. All patients will then receive as their initial analgesic oral acetaminophen 975 mg followed by morphine sulfate 0.05 mg/kg IV rounded to the nearest milligram.

E. Each patient will then be randomized in either of two arms:

1. Ultrasound guided serratus anterior plane block (SAPB) with 30mL 0.25% bupivacaine with epinephrine.
2. Ultrasound guided serratus anterior plane injection with placebo injection with 30mL of normal saline.

6. Investigators will be blinded to the arm that the patient has been randomized to, as the randomization will occur through the pharmacy dispensing the medication.

7. Using an online randomizer in blocks of 10, the pharmacy will dispense either 30mL of normal saline for the sham group, or 30mL of 0.25% bupivacaine with epinephrine for the nerve block group.

8. All patients will receive either SAPB or placebo injection within an hour of receiving the initial analgesics of acetaminophen and morphine.

9. If the patient still has a pain score ≥5 thirty minutes after the injection, the treating physician will be informed and the patient will be medicated at the treating physician's discretion.

10. The patient will be followed up with up to 24 hours throughout their hospital stay.

Data Collection Procedures:

A. Demographics 1. Age, sex, ethnicity, height B. Past medical history 1. Smoking status (current, prior, never smoker), diabetes, cirrhosis, chronic obstructive pulmonary disease (COPD), asthma, if patient uses home oxygen C. Injury Mechanism

1. Occupant in motor vehicle collision, fall from an elevation, fall down stairs, fall from standing, pedestrian or bicyclist struck by moving vehicle, bike collision or fall from bike while riding, driver or passenger in motorcycle/ATV/motorized scooter collision, assault, unknown mechanism, or other
2. Date and time of injury
3. GCS score
4. Injury Severity Scale D. Imaging

<!-- -->

1. Side of rib fractures
2. Number of rib fractures on x-ray and on CT chest
3. Rib fracture location: anterior, lateral, posterior, T1-12
4. Type of imaging showing rib fractures
5. Presence of following: atelectasis, hemothorax, infiltrate (right/left), interstitial edema, pneumothorax, pulmonary contusion E. Medication

1. Any medications type and dose given prior to randomization

F. At Time 0 (time of enrollment):

1. Vital signs
2. Resting pain score from 0-10
3. Deep breath pain score from 0-10
4. Slow Vital Capacity (SVC)

   a. Measured until 3 measurements are within 150mL of each other b. % predicted SVC is measured based on NHANES III Calculator using age, sex, ethnicity and height. If ethnicity not included in calculator will select Caucasian.

   c. Maximum SVC and maximum % predicted SVC
5. Symptoms after injection: sedation, dizziness, dysarthria, nausea, new cardiac rhythm (significant tachycardia or bradycardia, SVT, etc), new significantly increased shortness of breath, perioral numbness, pruritis, seizure, syncope, tinnitus, vomiting G. At Time 30 minutes post injection

<!-- -->

1. Vital signs
2. Resting pain score from 0-10
3. Deep breath pain score from 0-10
4. Slow Vital Capacity (SVC)

   1. Measured until 3 measurements are within 150mL of each other
   2. Percentage predicted SVC is measured based on NHANES III Calculator using age, sex, ethnicity and height. If ethnicity not included in calculator will select Caucasian.
   3. Maximum SVC and maximum % predicted SVC
5. Symptoms after injection: sedation, dizziness, dysarthria, nausea, new cardiac rhythm (significant tachycardia or bradycardia, SVT, etc), new significantly increased shortness of breath, perioral numbness, pruritis, seizure, syncope, tinnitus, vomiting H. At Time 60 minutes post injection

<!-- -->

1. Vital signs
2. Resting pain score from 0-10
3. Deep breath pain score from 0-10
4. Slow Vital Capacity (SVC)

<!-- -->

1. Measured until 3 measurements are within 150mL of each other
2. % predicted SVC is measured based on NHANES III Calculator using age, sex, ethnicity and height. If ethnicity not included in calculator will select Caucasian.
3. Maximum SVC and maximum % predicted SVC

5. Symptoms after injection: sedation, dizziness, dysarthria, nausea, new cardiac rhythm (significant tachycardia or bradycardia, SVT, etc), new significantly increased shortness of breath, perioral numbness, pruritis, seizure, syncope, tinnitus, vomiting I. At Time 3-6 hours post injection

1. Vital signs 2. Resting pain score from 0-10 3. Deep breath pain score from 0-10 4. Slow Vital Capacity (SVC)

1. Measured until 3 measurements are within 150mL of each other
2. % predicted SVC is measured based on NHANES III Calculator using age, sex, ethnicity and height. If ethnicity not included in calculator will select Caucasian.
3. Maximum SVC and maximum % predicted SVC 4. Symptoms after injection: sedation, dizziness, dysarthria, nausea, new cardiac rhythm (significant tachycardia or bradycardia, SVT, etc), new significantly increased shortness of breath, perioral numbness, pruritis, seizure, syncope, tinnitus, vomiting J. At Time 12 hours post injection 1. Vital signs 2. Resting pain score from 0-10 3. Deep breath pain score from 0-10 5. Slow Vital Capacity (SVC)

   1. Measured until 3 measurements are within 150mL of each other
   2. % predicted SVC is measured based on NHANES III Calculator using age, sex, ethnicity and height. If ethnicity not included in calculator will select Caucasian.
   3. Maximum SVC and maximum % predicted SVC

   5. Symptoms after injection: sedation, dizziness, dysarthria, nausea, new cardiac rhythm (significant tachycardia or bradycardia, SVT, etc), new significantly increased shortness of breath, perioral numbness, pruritis, seizure, syncope, tinnitus, vomiting J. On 24 hours post injection
   1. Vital signs
   2. Resting pain score from 0-10
   3. Deep breath pain score from 0-10
   4. Slow Vital Capacity (SVC)

<!-- -->

1. Measured until 3 measurements are within 150mL of each other
2. % predicted SVC is measured based on NHANES III Calculator using age, sex, ethnicity and height. If ethnicity not included in calculator will select Caucasian.
3. Maximum SVC and maximum % predicted SVC 5. Symptoms after injection: sedation, dizziness, dysarthria, nausea, new cardiac rhythm (significant tachycardia or bradycardia, SVT, etc), new significantly increased shortness of breath, perioral numbness, pruritis, seizure, syncope, tinnitus, vomiting K. Slow vital capacity

   1. Researchers will be trained on appropriate incentive spirometry technique by the respiratory therapy team and their accuracy will be confirmed 2. Patients will then be instructed to perform SVC, we will get 3 SVC measurements within 150mL of each other and then record the maximum SVC.

   3. Percent predicted vital capacity will be calculating using NHANES III L. Time to first rescue analgesia post injection M. Medications during first 24 hours of hospital stay

   1. 24 hour total morphine milligram equivalent consumption

   1. Calculated based on CDC Morphine Milligram Equivalence (MME) Calculator: https://www.cdc.gov/drugoverdose/prescribing/app.html 2. Any antemetics used after injection within 24 hours after enrollment 3. Time to administration of first rescue analgesia post injection N. Nerve Block performed during inpatient stay

   1. List date/time/type of any additional nerve blocks performed for rib fracture pain after the study injection during the patient's hospital stay

   O. Pulmonary complications:

   1. New O2 requirement, BIPAP or intubation, transfer to ICU for respiratory issue, development of pneumonia, readmission for pulmonary issue, new need for home O2 P. Nerve Block Complications

   1. Development of cellulitis at site of block during hospital stay 2. Pneumothorax occurring within 12 hours of injection Q. Discharge Data
   1. If cellulitis developed at the site of injection during hospital stay
   2. If a pneumothorax on the same side of the injection occurred within 12 hours of block R. Imaging

   1. Videos of the nerve block performance will be recorded in each patient. These images will later be de-identified and reviewed by two independent reviewers not involved in the study to determine visually whether the planar spread of anesthetic was correctly placed or not correctly placed.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Presumed/Clinically apparent 2 or more acute unilateral rib fractures between T3-T9
3. Pain Score 5 or greater

Exclusion Criteria:

1. GCS<13
2. Penetrating trauma
3. Pregnant
4. Unable to give consent due to dementia or altered mental status
5. Unable to perform spirometry
6. Requiring immediate surgical intervention
7. Known allergy to amide-type local anesthetics
8. Signs of infection or laceration at injection site
9. Systolic BP <100 mmHg
10. History of chronic pain, chronic use of analgesics
11. History of substance abuse
12. Painful distracting injury (injury causing significant pain that distracts the patient from having reliable scoring of rib fracture pain, i.e. femur fracture, dislocated joint)
13. If patient received any other pain medication besides ketamine prior to the block
14. Only posterior rib fractures present
15. known allergy to acetaminophen
16. Known allergy to morphine sulfate

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Lin, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placeoo Injection Group: The injection of normal saline into the chest muscle is performed with an ultrasound machine which can see the needle as it enters the muscle. The skin is cleaned with a sterile solution and the needle is guided right next to the chest muscle where saline is injected. After the injection, the needle is taken out.
  Acetaminophen: receive ketamine 0.15 mg/kg IV in 100 mL normal saline over 30 minutes for pain
  Saline: The injection of saline into the chest muscle is performed with an ultrasound machine which can see the needle as it enters the muscle.
Period: Overall Study
Arm/Group | Serratus Anterior Plane Block Group | Placeoo Injection Group
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Serratus Anterior Plane Block Group | Placeoo Injection Group | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Pain Control
Description: Pain score on 11 point Numeric Rating Scale ranging 0-10 with 0 being no pain, 5 being moderate pain, and 10 being very severe pain
Time Frame: 60 minutes
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Serratus Anterior Plane Block Group | Placeoo Injection Group
Number analyzed (Participants) | 1 | 2
score on a scale | 5 [5 to 5] | 2.5 [0 to 5]

ADVERSE EVENTS:
Time Frame: 60 minutes
Arm/Group | Serratus Anterior Plane Block Group | Placeoo Injection Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT04530149/Prot_SAP_001.pdf